CLINICAL TRIAL: NCT03143686
Title: ACURATE TA™ Valve Implantation: SAVI Registry (Surveillance Plan #2011-02) (TA-SAVI)
Status: Completed | Type: Observational
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Other Study IDs: 2011-02
Record Dates: First submitted 2014-12-08; First posted 2017-05-08 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: Severe symptomatic Aortic Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACURATE TA™ Transapical Aortic Bioprosthesis: The first two hundred and fifty (250) patients in whom the commercial, or CE Mark, ACURATE TATM Transapical Aortic Bioprosthesis is implanted.
  Interventions: Device: ACURATE TA™ Transapical Aortic Bioprosthesis

INTERVENTIONS:
Device: ACURATE TA™ Transapical Aortic Bioprosthesis — ACURATE TA™ Transapical Aortic Bioprosthesis is intended for subjects with severe symptomatic aortic stenosis and are considered high risk for surgical conventional Aortic Valve Replacement.
  Other Names: ACURATE TA™ Transapical Aortic Bioprosthesis and delivery System

SUMMARY:
Post-market registry on ACURATE TA™ Transapical Aortic Bioprosthesis and ACURATE TA™ Delivery System implantation in patients presenting severe symptomatic aortic stenosis to provide safety surveillance of the device.

DETAILED DESCRIPTION:
A single arm, prospective, multicenter, non-randomized and open registry up to 1 Year Follow-up with the Symetis ACURATE TA™ which is an aortic bioprosthesis for minimal invasive implantation via transapical access to treat patients with severe symptomatic aortic stenosis where surgical aortic valve replacement (SAVR) via open surgery is considered to be associated with high surgical risk for evaluating the safety and performance of the implantation and the safety at 30-Day Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient has severe aortic stenosis
* Native aortic annulus diameter from ≥ 21mm up to ≤ 27mm
* Patient willing to participate in the study and provides signed EC-approved informed consent
* The subject and treating physician agree the subject will return for all required post-procedure follow-up visits

Exclusion Criteria:

* Patients are excluded from the registry if they are not eligible for transcatheter treatment of severe aortic stenosis with the ACURATE TA™ and Delivery System as per the Instructions For Use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ACURATE TA™ is approved for use to treat patients with severe aortic stenosis. The registry includes all comer patients following the Instructions For Use.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Rate of major cardiac and cerebrovascular event (MACCE) at 30 days and at 12 months post-implant | 30 days and 12 Months Follow-up
  Rate of major cardiac and cerebrovascular event (MACCE) at 30 days and at 12 months post-implant .
  MACCE defined as All cause mortality, Re-intervention, Myocardial Infarction, or Stroke.

SECONDARY OUTCOMES:
Procedural Success post-implantation (up to 24 hours after device implantation) | Post-Implantation (up to 24 hours after device implantation)
  Procedural success defined as successful ACURATE TA™ implantation at intended site and adequate device functioning immediately post-implantation and without intra-procedural mortality
Device success at 30 days and 12 Months follow-up | 30 days and 12 Months follow-up
  Device success at 30 day and 12 month follow-up visit defined as adequate functioning of the ACURATE TA™ as confirmed by echocardiography.

CONTACTS AND LOCATIONS:
Locations (17):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Germany (14):
  - RWTH Aachen, Aachen
  - Zentralklinik Bad Berka, Bad Berka
  - Kerckhoff Klinik Bad Nauheim, Bad Nauheim
  - Herz-und Gefäss-Klinik GmbH, Bad Neustadt an der Saale
  - Schüchtermann-Schiller'sche Kliniken GmbH, Bad Rothenfelde
  - Uniklinik Köln Herzzentrum, Cologne
  - Herzzentrum Dresden Universitätsklinik, Dresden
  - Klinik für Tgorax und Gefässchirurgie, Essen
  - Universitäres Herzzentrum, Hamburg
  - Klinik für Herzchirurgie, Karlsruhe
  - Herzzentrum Leipzig, Leipzig
  - Universitäts Medizin Mainz, Mainz
  - Universitätsklinikum Regensburg, Regensburg
  - Sana Herzchirurgie Stuttgart GmbH, Stuttgart
- Policlinico s. Orsola-Malpighi, Bologna, Italy
- Inselspital-Stiftung, Bern, Switzerland